CLINICAL TRIAL: NCT04872725
Title: The Effect of Covid-19 Process on Time Management, Participation and Leisure Activity
Brief Title: The Effect of Covid-19 Process
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, mbudak, Principal Investigator, Medipol University
Other Study IDs: Covid-19 OT
Record Dates: First submitted 2021-05-02; First posted 2021-05-04 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Covid19; Participation, Patient
Keywords: Covid-19; leisure time activities; participation; time management
MeSH Terms: conditions — COVID-19; Patient Participation | interventions — Time Management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Time management & participation & the leisure time activity — evaluated in terms of leisure time activities, time management and participation

SUMMARY:
Objective: The purpose of this study was to investigate the effect of the Covid-19 process on time management, participation, and leisure time activity.

Methods: 531 individuals aged between 18-65 were included in the study. The individuals were evaluated with the Assessment Of Time Management Skills (ATMS) in terms of time management, with the Social Isolation Questionnaire (SIQ) in terms of participation, and with the Interest Checklist (IC) in terms of leisure time activities.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18-65
* lived the Covid-19 process in Turkey

Exclusion Criteria:

* did not complete the scales
* did not live in Turkey

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: aged between 18-65, signed "Informed Consent Form" and fulfilled the inclusion criteria
Sampling Method: Probability Sample
Enrollment: 531 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Assessment of Time Management Skills | from March to June
  It is a 30-item assessment tool that describes how different practical situations related to time management in a person's life are resolved or one's possible views on one's own time management skills. The scale is in 4-likert format and is evaluated as "1: Never, 2: Sometimes, 3: Most of the time, 4: Always" and the scores obtained are scored between 30-120. High scores indicate that time management skills and practices perform better. Eight items are reverse scored (items 7, 9, 10, 12, 18, 23, 26 and 30)
Social Isolation Questionnaire | from March to June
  It consists of 6 items that evaluate the loneliness and perceived social isolation of the individual. A minimum score of 0 and a maximum of 24 points are obtained on the scale. 0 points means total social isolation, 24 points means high social relations. A value between 0-10 means complete social isolation, a value between 12-15 means isolation, a value between 16-18 means partial isolation, a value between 19-21 means social relation, and a value between 21-24 means a high social relationship.
Interest Checklist | from March to June
  It is suitable for all population groups. The areas of interest are divided into 9 categories in each section, where relevant activities are listed and the individual can add their own activity. For each activity, it questions participation in the activity (in the past, ongoing and / or planned in the future) and degree of interest (strong, little, nothing).

CONTACTS AND LOCATIONS:
Overall Officials: Miray BUDAK, PhD, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Beykoz, Istanbul, Turkey (Türkiye)